CLINICAL TRIAL: NCT02926833
Title: A Phase 1-2 Multi-Center Study Evaluating the Safety and Efficacy of KTE-C19 in Combination With Atezolizumab in Subjects With Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Study of Safety and Efficacy of KTE-C19 in Combination With Atezolizumab in Adults With Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Acronym: ZUMA-6
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-106
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Refractory Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — axicabtagene ciloleucel; atezolizumab; Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: This study uses a single group design. The arms reported in the Arms and Intervention section are based on the atezolizumab dosing schedule in the 4 Cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 Cohort 1: KTE-C19 + ATZ (After 21 Days of KTE-C19) (Experimental): Participants received conditioning chemotherapy consisting of 30 mg/m^2 fludarabine and 500 mg/m^2 cyclophosphamide intravenous (IV) infusion per day for 3 days followed by KTE-C19 IV infusion at a target dose of 2 x 10^6 anti-CD19 chimeric antigen receptor (CAR) T cells/kg followed by 4 doses of atezolizumab (ATZ) (1200 mg/dose) IV infusion every 21 days, beginning 21 days following KTE-C19.
  Interventions: Biological: KTE-C19; Biological: Atezolizumab; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 1 Cohort 2: KTE-C19 + ATZ (After 14 Days of KTE-C19) (Experimental): Participants received conditioning chemotherapy consisting of 30 mg/m^2 fludarabine and 500 mg/m^2 cyclophosphamide IV infusion per day for 3 days followed by KTE-C19 IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg followed by 4 doses of ATZ (1200 mg/dose) IV infusion every 21 days, beginning 14 days following KTE-C19.
  Interventions: Biological: KTE-C19; Biological: Atezolizumab; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 1 Cohort 3: KTE-C19 + ATZ (After 1 Day of KTE-C19) (Experimental): Participants received conditioning chemotherapy consisting of 30 mg/m^2 fludarabine and 500 mg/m^2 cyclophosphamide IV infusion per day for 3 days followed by KTE-C19 IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg followed by 4 doses of ATZ (1200 mg/dose) IV infusion every 21 days, beginning 1 day following KTE-C19.
  Interventions: Biological: KTE-C19; Biological: Atezolizumab; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 2: KTE-C19 + ATZ (After 1 Day of KTE-C19) (Experimental): Participants received conditioning chemotherapy consisting of 30 mg/m^2 fludarabine and 500 mg/m^2 cyclophosphamide IV infusion per day for 3 days followed by KTE-C19 IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg followed by 4 doses of ATZ (1200 mg/dose) IV infusion every 21 days, beginning 1 day following KTE-C19.
  Interventions: Biological: KTE-C19; Biological: Atezolizumab; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: KTE-C19 — A single infusion of KTE-C19 CAR-T cells administered intravenously
  Other Names: Axicabtagene ciloleucel; Yescarta®
Biological: Atezolizumab — Administered intravenously
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously

SUMMARY:
The primary objective of phase 1 is to evaluate the safety of KTE-C19 and atezolizumab combination regimens.

The primary objective of phase 2 is to evaluate the efficacy of KTE-C19 and atezolizumab, as measured by complete response rate in participants with refractory diffuse large B-cell lymphoma (DLBCL).

Participants who received an infusion of KTE-C19 will complete the remainder of the 15 year follow-up assessments in a separate long-term follow-up study, KT-US-982-5968 (NCT05041309).

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed DLBCL
2. Chemotherapy-refractory disease, defined as one or more of the following:

   * Stable disease (duration of stable disease must be less than or equal to 6 months) or progressive disease as best response to most recent chemotherapy containing regimen
   * Disease progression or recurrence less than or equal to 12 months of prior autologous stem cell transplantation (SCT)
3. Individuals must have received adequate prior therapy including at a minimum:

   * Anti-cluster of differentiate 20 (anti-CD20) monoclonal antibody unless investigator determines that tumor is CD20-negative; and
   * an anthracycline containing chemotherapy regimen
4. At least one measurable lesion per revised International Working Group (IWG) Response Criteria
5. Age 18 years or older
6. Eastern cooperative oncology group (ECOG) performance status of 0 or 1
7. Adequate organ and bone marrow function
8. All individuals or legally appointed representatives/caregivers, must personally sign and date the institutional review board (IRB)/independent ethics committee (IEC) approved consent form before initiating any study specific procedures or activities.

Key Exclusion Criteria:

1. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g., cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years
2. History of allogeneic stem cell transplantation
3. Prior CAR therapy or other genetically modified T cell therapy
4. Clinically significant active infection
5. Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive)
6. Individuals with detectable cerebrospinal fluid malignant cells or brain metastases or with a history of cerebrospinal fluid malignant cells or brain metastases
7. History of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with central nervous system (CNS) involvement
8. History of autoimmune disease. Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and participants with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study.
9. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computed tomography (CT) scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
10. Prior treatment with Programmed Cell Death Ligand 1 (PD-L1) inhibitor, PD-1 inhibitor, anti-CTLA4, anti-CD137, anti-OX40 or other immune checkpoint blockade or activator therapy with the exception of Individuals who received atezolizumab in this study and are eligible for re-treatment
11. Prior CD19 targeted therapy

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Stanford Cancer Center, Palo Alto, California
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Background] Jacobson CA, Locke FL, Miklos DB, Herrera AF, Westin JR, Lee J, et al. End of Phase 1 results for ZUMA-6: Axicabtagene ciloleucel (axi-cel) in combination with atezolizumab for the treatment of patients with refractory diffuse large B cell lymphoma. Presented at ASH, 2018.
- [Background] Locke FL, Westin JR, Miklos DB, Herrera AF, Jacobson CA, Lee J, et al. Phase 1 results from ZUMA-6: Axicabtagene ciloleucel (axi-cel; KTE-C19) in combination with atezolizumab for the treatment of patients with refractory diffuse large B cell lymphoma. Presented at ASH, 2018, presentation #2628.
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 44 participants were screened.
Groups:
- Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19): Participants received conditioning chemotherapy consisting of 30 mg/m^2 fludarabine and 500 mg/m^2 cyclophosphamide intravenous (IV) infusion per day for 3 days followed by KTE-C19 IV infusion at a target dose of 2 x 10^6 anti-CD19 chimeric antigen receptor (CAR) T cells/kg followed by 4 doses of atezolizumab (ATZ) (1200 mg/dose) IV infusion every 21 days, beginning 21 days following KTE-C19.
- Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19): Participants received conditioning chemotherapy consisting of 30 mg/m^2 fludarabine and 500 mg/m^2 cyclophosphamide IV infusion per day for 3 days followed by KTE-C19 IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg followed by 4 doses of ATZ (1200 mg/dose) IV infusion every 21 days, beginning 14 days following KTE-C19.
- Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19); Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19): Participants received conditioning chemotherapy consisting of 30 mg/m^2 fludarabine and 500 mg/m^2 cyclophosphamide IV infusion per day for 3 days followed by KTE-C19 IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg followed by 4 doses of ATZ (1200 mg/dose) IV infusion every 21 days, beginning 1 day following KTE-C19.
Period: Overall Study
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Started | 3 | 4 | 7 | 23
Completed | 1 | 0 | 1 | 0
Not Completed | 2 | 4 | 6 | 23
Not completed — Death | 1 | 1 | 2 | 13
Not completed — Lost to Follow-up | 1 | 2 | 0 | 3
Not completed — Full Consent Withdrawal | 0 | 0 | 0 | 2
Not completed — Rolled Over to Long-term Follow-up Study | 0 | 0 | 3 | 4
Not completed — Investigator Decision | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Partial Withdrawal of Consent | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants treated with any dose of KTE-C19.
Groups:
- Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19): Participants received conditioning chemotherapy consisting of 30 mg/m^2 fludarabine and 500 mg/m^2 cyclophosphamide IV infusion per day for 3 days followed by KTE-C19 IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg followed by 4 doses of ATZ (1200 mg/dose) IV infusion every 21 days, beginning 21 days following KTE-C19.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 22 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 6 | 18 | 28
  >=65 years | 1 | 1 | 0 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (14.80) | 42.7 (19.50) | 53.2 (6.18) | 58.4 (7.40) | 56 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 4 | 8 | 14
  Male | 3 | 1 | 2 | 14 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 2 | 2 | 6 | 20 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1 | 3 | 5
  White | 2 | 3 | 5 | 18 | 28
  Other | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6 | 22 | 34

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as the following KTE-C19-related or ATZ-related events with an onset from immediately after the first ATZ infusion through 21 days after the first ATZ infusion: Grade 4 hematologic toxicity lasting > 30 days (except lymphopenia or B-cell aplasia); All KTE-C19- or ATZ-related Grade 3 non-hematologic toxicities lasting for > 7 days and all KTE-C19- or ATZ-related Grade 4 non-hematologic toxicities regardless of duration.
Time Frame: Baseline up to 21 days
Population: DLT Evaluable Set included all participants in Phase 1 treated with KTE-C19 and at least 1 dose of ATZ who either received target KTE-C19 dose and followed for at least 21 days after first ATZ infusion; or received a dose of KTE-C19 lower than target for that cohort and a subsequent ATZ infusion and experienced a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 1

2. Primary Outcome: Phase 1 and 2: Complete Response Rate (CRR)
Description: CRR was assessed based on the International Working Group Revised Response Criteria for Malignant Lymphoma (Cheson, 2007), and was defined as the percentage of participants achieving a complete response (CR) as assessed by the study investigators. CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease.
Time Frame: From enrollment until first occurrence of CR or PR (maximum duration: 6.2 years)
Population: The Modified Intent-to-Treat Analysis (mITT) Set included all participants enrolled in Phase 1 Cohort 3 and Phase 2 and treated with target dose of KTE-C19 and at least one dose of atezolizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ: Participants received conditioning chemotherapy consisting of 30 mg/m^2 fludarabine and 500 mg/m^2 cyclophosphamide IV infusion per day for 3 days followed by KTE-C19 IV infusion at a target dose of 2 x 10^6 anti-CD19 CAR T cells/kg followed by 4 doses of ATZ (1200 mg/dose) IV infusion every 21 days, beginning 1 day following KTE-C19.
Arm/Group | Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ
Number analyzed (Participants) | 28
percentage of participants | 54 [34 to 72]

3. Secondary Outcome: Phase 1 and 2: Objective Response Rate (ORR)
Description: ORR was assessed based on the International Working Group Revised Response Criteria for Malignant Lymphoma (Cheson, 2007), and was defined as the percentage of participants achieving a CR or partial response (PR) as assessed by the study investigators. CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. PR was defined at least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses. Participants who did not meet the criteria for objective response by the analysis cutoff date were considered non-responders.
Time Frame: From enrollment until first occurrence of CR or PR (maximum duration: 6.2 years)
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ
Number analyzed (Participants) | 28
percentage of participants | 75 [55 to 89]

4. Secondary Outcome: Phase 1 and 2: Duration of Response (DOR)
Description: DOR for participants who experienced an objective response was defined as the date of their first confirmed objective response (CR or PR) to disease progression per the revised International Working Group Response Criteria for Malignant Lymphoma (Cheson, 2007) or death regardless of cause. CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. PR was defined at least a 50% decrease in SPD of up to six of the largest dominant nodes or nodal masses. Disease progression was defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir. The Kaplan-Meier approach was used to estimate DOR.
Time Frame: From the date of first confirmed objective response (CR or PR) to disease progression or death regardless of cause (maximum duration: 6.2 years)
Population: Participants in the mITT Analysis Set with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ
Number analyzed (Participants) | 21
months | 41.4 [1.8 to NA] — Due to less number of participants with an event, upper limit of 95% confidence interval (CI) was not estimable.

5. Secondary Outcome: Phase 1 and 2: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the KTE-C19 infusion date to the date of disease progression per the revised International Working Group Response Criteria for Malignant Lymphoma (Cheson, 2007) or death from any cause. Disease progression was defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir. The Kaplan-Meier approach was used to estimate PFS.
Time Frame: From the date of first KTE-C19 infusion to disease progression or death regardless of cause (maximum duration: 6.2 years)
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ
Number analyzed (Participants) | 28
months | 9 [3.1 to NA] — Due to less number of participants with an event, upper limit of 95% CI was not estimable.

6. Secondary Outcome: Phase 1 and 2: Overall Survival (OS)
Description: OS was defined as the time from KTE-C19 infusion to the date of death from any cause. The Kaplan-Meier approach was used to estimate OS.
Time Frame: From the date of first KTE-C19 infusion to the date of death regardless of cause (maximum duration: 6.2 years)
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ
Number analyzed (Participants) | 28
months | 32.2 [11.6 to NA] — Due to less number of participants with an event, upper limit of 95% CI were not estimable.

7. Secondary Outcome: Phase 1 and 2: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event was defined as any untoward medical occurrence in a clinical trial participant. The event did not necessarily have a relationship with study treatment. Adverse events included worsening of a pre-existing medical condition. Worsening indicated that the pre-existing medical condition had increased in severity, frequency, and/or duration or had an association with a worse outcome. A pre-existing condition that had not worsened during the study or involved an intervention such as elective cosmetic surgery or a medical procedure while in study, was not considered an adverse event. TEAEs included all AEs with onset on or after initiation of axicabtagene ciloleucel.
Time Frame: Up to 1.8 years
Population: The Safety Analysis Set was defined as all participants treated with any dose of KTE-C19.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6 | 22
percentage of participants | 100 | 100 | 100 | 100

8. Secondary Outcome: Phase 1 and 2: Percentage of Participants With Serum Chemistry Toxicity Grade Shifts to Grade 3 or Higher Resulting From Increased Parameter Values
Description: Post axicabtagene ciloleucel infusion lab toxicities were reported. It included lab toxicities observed on or after the axicabtagene ciloleucel infusion date.
  ALT = alanine aminotransferase; ALP = alkaline phosphatase; AST = aspartate aminotransferase.
Time Frame: Up to 1.8 years
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6 | 22
percentage of participants
  Shift to Grade 3 ALT | 0 | 0 | 0 | 5
  Shift to Grade 4 ALT | 0 | 0 | 0 | 5
  Shift to Grade 3 ALP | 0 | 0 | 0 | 14
  Shift to Grade 3 AST | 0 | 0 | 0 | 9
  Shift to Grade 4 AST | 0 | 0 | 0 | 5
  Shift to Grade 3 bilirubin | 0 | 0 | 0 | 9
  Shift to Grade 4 calcium | 0 | 0 | 0 | 5
  Shift to Grade 3 creatinine | 0 | 0 | 0 | 9
  Shift to Grade 4 creatinine | 0 | 0 | 0 | 5
  Shift to Grade 3 direct bilirubin | 33 | 33 | 17 | 14
  Shift to Grade 3 glucose | 0 | 0 | 0 | 18
  Shift to Grade 4 glucose | 0 | 0 | 0 | 14

9. Secondary Outcome: Phase 1 and 2: Percentage of Participants With Serum Chemistry Toxicity Grade Shifts to Grade 3 or Higher Resulting From Decreased Parameter Values
Description: Post axicabtagene ciloleucel infusion lab toxicities were reported. It included lab toxicities observed on or after the axicabtagene ciloleucel infusion date.
Time Frame: Up to 1.8 years
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6 | 22
percentage of participants
  Shift to Grade 3 albumin | 33 | 0 | 0 | 9
  Shift to Grade 3 calcium | 33 | 0 | 0 | 5
  Shift to Grade 4 calcium | 0 | 0 | 0 | 18
  Shift to Grade 3 phosphate | 67 | 67 | 33 | 36
  Shift to Grade 4 phosphate | 0 | 0 | 0 | 36
  Shift to Grade 3 potassium | 0 | 0 | 0 | 14
  Shift to Grade 3 sodium | 67 | 0 | 17 | 14
  Shift to Grade 4 glucose | 0 | 0 | 17 | 0

10. Secondary Outcome: Phase 1 and 2: Percentage of Participants With Hematology Toxicity Grade Shifts to Grade 3 or Higher Resulting From Increased Parameter Values
Description: as for outcome 9
Time Frame: Up to 1.8 years
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6 | 22
percentage of participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Phase 1 and 2: Percentage of Participants With Hematology Toxicity Grade Shifts to Grade 3 or Higher Resulting From Decreased Parameter Values
Description: as for outcome 9
Time Frame: Up to 1.8 years
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6 | 22
percentage of participants
  Shift to Grade 3 hemoglobin | 100 | 67 | 83 | 59
  Shift to Grade 3 leukocytes | 0 | 0 | 33 | 18
  Shift to Grade 4 leukocytes | 100 | 100 | 67 | 77
  Shift to Grade 4 lymphocytes | 100 | 100 | 100 | 86
  Shift to Grade 3 neutrophils | 0 | 33 | 17 | 14
  Shift to Grade 4 neutrophils | 100 | 67 | 83 | 73
  Shift to Grade 3 platelets | 33 | 0 | 17 | 18
  Shift to Grade 4 platelets | 33 | 67 | 17 | 32

12. Secondary Outcome: Phase 1 and 2: Peak Anti-CD19 CAR T-Cell (KTE-C19) Level (Maximum Observed Plasma Concentration) in Blood
Time Frame: Pre-infusion (Baseline); Post-infusion: Days 7 (Phase 2), 14, 22 (Phase 2), 28 (Phase 2; optional), 35 (Phase 1, Cohort 3; optional), 43, 49 (optional), 64, 69 (optional), 94; long-term follow-up: every 3 months from Month 6 to Month 18, and Month 24
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6 | 22
cells/μL | 86.87 (67.17) | 167.88 (91.58) | 60.71 (70.66) | 60.22 (60.24)

13. Secondary Outcome: Phase 1 and 2: Percentage of Participants With Anti-KTE-C19 Antibodies
Time Frame: Baseline (pre-conditioning chemotherapy); Day 0 (pre-KTE-C19 infusion); Days 1, 4, 7, 14, 22 , 28, Day 35, 49, 69, and 94 post-KTE-C19 infusion
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6 | 22
percentage of participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Phase 1 and 2: Atezolizumab Levels in Blood
Time Frame: Days 1, 14, 21, 22, 35, 42, 43, 56, 63, 64, 77, 84, 154, and 174
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6 | 22
ng/mL
  Day 1: number analyzed (Participants) | 0 | 0 | 6 | 19
  Day 1 |  |  | 373000 (65300) | 328000 (89100)
  Day 14: number analyzed (Participants) | 0 | 3 | 0 | 0
  Day 14 |  | 435000 (61500) |  |
  Day 21: number analyzed (Participants) | 3 | 0 | 0 | 0
  Day 21 | 403000 (46100) |  |  |
  Day 22: number analyzed (Participants) | 0 | 0 | 4 | 17
  Day 22 |  |  | 73900 (27900) | 110000 (126000)
  Day 35: number analyzed (Participants) | 0 | 3 | 0 | 0
  Day 35 |  | 84200 (14300) |  |
  Day 42: number analyzed (Participants) | 3 | 0 | 0 | 0
  Day 42 | 98800 (16500) |  |  |
  Day 43: number analyzed (Participants) | 0 | 0 | 4 | 15
  Day 43 |  |  | 138000 (78700) | 136000 (69900)
  Day 56: number analyzed (Participants) | 0 | 2 | 0 | 0
  Day 56 |  | 176000 (2828.43) |  |
  Day 63: number analyzed (Participants) | 3 | 0 | 0 | 0
  Day 63 | 175000 (7505.55) |  |  |
  Day 64: number analyzed (Participants) | 0 | 0 | 5 | 14
  Day 64 |  |  | 159000 (91600) | 185000 (88700)
  Day 77: number analyzed (Participants) | 0 | 3 | 0 | 0
  Day 77 |  | 240000 (33000) |  |
  Day 84: number analyzed (Participants) | 3 | 0 | 0 | 0
  Day 84 | 209000 (24800) |  |  |
  Day 154: number analyzed (Participants) | 0 | 0 | 1 | 3
  Day 154 |  |  | 13600 | 66800 (58900)
  Day 174: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 174 | 91000 |  |  |

15. Secondary Outcome: Phase 1 and 2: Percentage of Participants With Anti-Atezolizumab Antibodies
Time Frame: as for outcome 13
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
Number analyzed (Participants) | 3 | 3 | 6 | 22
percentage of participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Phase 1 and 2: Peak Serum Levels of C-Reactive Protein (CRP) in Blood
Time Frame: Baseline (pre-conditioning chemotherapy); Day 0 (pre-KTE-C19 infusion); Days 1, 4, 7, and 14, and 22 , optional Day 28 (Phase 2) or Day 35 (Phase 1 Cohort 3), optional Day 49, optional Day 69, and Day 94 post-KTE-C19 infusion
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ
Number analyzed (Participants) | 28
mg/L | 174.03 [51.78 to 496.00]

17. Secondary Outcome: Phase 1 and 2: Peak Serum Levels of C-X-C Motif Chemokine 10 (CXCL10), Interferon-Gamma (IFN-γ), Interleukin-1 Receptor Antagonist (IL-1RA), Interleukin (IL)-2, IL-6, IL-8, IL-15, and Tumor Necrosis Factor-Alpha (TNF-α) in Blood
Time Frame: as for outcome 16
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ
Number analyzed (Participants) | 28
pg/mL
  CXCL 10 | 2000.00 [444.80 to 2000.00]
  IFN-γ | 587.80 [15.60 to 1876.00]
  IL-1RA | 2469.60 [541.40 to 9000.00]
  IL-2 | 17.55 [1.80 to 152.70]
  IL-6 | 121.55 [4.30 to 976.00]
  IL-8 | 180.65 [18.60 to 750.00]
  IL-15 | 48.95 [19.10 to 161.20]
  TNF-α | 8.20 [3.40 to 55.50]

18. Secondary Outcome: Phase 1 and 2: Peak Serum Levels of Ferritin in Blood
Time Frame: as for outcome 16
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ
Number analyzed (Participants) | 28
ng/mL | 1427.39 [219.92 to 23100]

19. Secondary Outcome: Phase 1 and 2: Peak Serum Levels of Interleukin-2 Receptor Alpha (IL-2Rα) in Blood
Time Frame: as for outcome 16
Population: Participants in the mITT Analysis Set were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Phase 1 (Cohort 3) + Phase 2: KTE-C19 + ATZ
Number analyzed (Participants) | 28
ng/mL | 17.75 [3.45 to 57.77]

ADVERSE EVENTS:
Time Frame: Adverse Events: Up to 1.8 years; All-Cause Mortality: Enrollment up to 30 days after completion of the final dose of atezolizumab, or 24 months after the KTE-C19 infusion or until disease progression, whichever was longer (maximum duration: 6.2 years)
Description: All-Cause Mortality: Participants from All Enrolled Analysis Set were included.
  Serious Adverse Events and Other Adverse Events: The Safety Analysis Set was defined as all participants treated with any dose of KTE-C19.
Arm/Group | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19)
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/4 | 2/7 | 14/23
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/6 | 15/22
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) (N=3) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) (N=3) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) (N=6) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19) (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Jejunal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 3
Swelling face (General disorders) | 0 | 0 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 1 | 1 | 4
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 0 | 2
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1: KTE-C19 + ATZ (21 Days After KTE-C19) (N=3) | Phase 1 Cohort 2: KTE-C19 + ATZ (14 Days After KTE-C19) (N=3) | Phase 1 Cohort 3: KTE-C19 + ATZ (1 Day After KTE-C19) (N=6) | Phase 2: KTE-C19 + ATZ (1 Day After KTE-C19) (N=22)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 4 | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 4 | 10
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 8
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Ear pruritus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 11
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 5 | 8
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 5
Application site paraesthesia (General disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 1 | 10
Fatigue (General disorders) | 2 | 3 | 4 | 11
Gait disturbance (General disorders) | 0 | 0 | 0 | 5
Malaise (General disorders) | 0 | 1 | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 2
Oedema (General disorders) | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 3 | 3 | 6 | 21
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 3
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1 | 2
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 1 | 0
Dacryocystitis (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal infection (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 3
Parotitis (Infections and infestations) | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0
Immunoglobulins decreased (Investigations) | 1 | 0 | 0 | 0
Interleukin level increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 2 | 10
Platelet count decreased (Investigations) | 1 | 0 | 2 | 7
Weight decreased (Investigations) | 1 | 2 | 0 | 2
Weight increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 5
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 1 | 1 | 3
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 4
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 3
Encephalopathy (Nervous system disorders) | 3 | 1 | 2 | 7
Headache (Nervous system disorders) | 1 | 1 | 4 | 13
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 2 | 2 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 4
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 6
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1 | 3
Hypotension (Vascular disorders) | 3 | 2 | 4 | 9
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Amendment 1 (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT02926833/Prot_000.pdf
  • Study Protocol: Amendment 2 (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT02926833/Prot_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan: Original (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT02926833/SAP_003.pdf
  • Statistical Analysis Plan: Supplemental Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT02926833/SAP_004.pdf